CLINICAL TRIAL: NCT05450263
Title: Preventing Chronicity of Sub-acute Low Back Pain by Altering the Neural Emotional Response to Pain - a Pilot Study Addressing the Efficacy and Feasibility of an Interoceptive Exposure Technique.
Brief Title: Preventing Chronicity of Sub-acute Low Back Pain by Altering the Neural Emotional Response to Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to recruit participants for this study.
Sponsor: Orton Orthopaedic Hospital (Other)
Responsible Party: Principal Investigator, Leena Ristolainen, Tage Orenius, Clinical psychologist, Principal Investigatior, tage.orenius@orton.fi, Leena Ristolainen as a co-author. This registration was submitted together with Tage Orenius, Orton Orthopaedic Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Research Institute Orton
Record Dates: First submitted 2022-06-22; First posted 2022-07-08 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Preventive Medicine
Keywords: prevention; sub-acute; low back pain; interoceptive
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sub-acute low back pain active intervention (Active Comparator): To assess the efficacy of IET on the chronification of LBP, participants who are found to have a higher risk of pain chronification due to the presence of a biomarker (positive mPFC-Nac connectivity) will be randomized to the intervention group (IET)
  Interventions: Behavioral: Interoceptive exposure
- Sub-acute low back pain passive intervention (Sham Comparator): Control group, treatment as usual.
  Interventions: Behavioral: Interoceptive exposure
- No intervention (No Intervention)

INTERVENTIONS:
Behavioral: Interoceptive exposure — A pilot study addressing the efficacy and feasibility of an interoceptive exposure technique.
  Arms: Sub-acute low back pain active intervention; Sub-acute low back pain passive intervention

SUMMARY:
Aim of the study It could be stated that chronification of low back pain in some respects depends on the emotional reactions to the acute pain state. This approach enables advancing novel therapeutics for preventing pain chronification by altering the pain-related affective states. At present, no publication evaluating the efficacy of IET in altering brain responses related to sub-acute low back pain seems available. Neither have we found any studies specifically addressing the efficacy of mindfulness training on the functional connection between PFC and NAc.

The aim of this study project is three-fold:

1. A systematic literature review of behavioural methods in the prevention of low back pain chronicity Orenius T, Silén E, Nuortimo A, Ristolainen L. Psychological interventions in preventing chronicity of sub-acute back pain: a systematic review. Scand J Pain. 2022 Jan 24;22(2):211-217. doi: 10.1515/sjpain-2021-0063. PROSPERO: CRD42019053580
2. A pilot study (n=7+7) to address the efficacy and feasibility of IET in preventing chronicity of sub-acute pain
3. A full scale study (n=20+20) addressing the efficacy and feasibility of IET in the prevention of chronicity of sub-acute low back pain

DETAILED DESCRIPTION:
To assess the efficacy of IET on the chronification of LBP, participants who are found to have a higher risk of pain chronification due to the presence of a biomarker (positive mPFC-Nac connectivity) will be randomized to the intervention group (IET) or control group A (treatment as usual). To assess how well this biomarker predicts the chronification of LBP, participants who are not found to have the biomarker will be assigned to control group B (treatment as usual).

ELIGIBILITY:
Inclusion Criteria:

The selection of subjects will meet same criteria as in the study by Baliki et al. (2010).

* Low back pain diagnosed by a clinician
* Low back pain intensity > 40/100 on NRS
* Low back pain duration 4-12 weeks

Exclusion Criteria:

* Other chronic painful condition
* Systemic disease
* History of head injury
* Diagnosed psychiatric disorders
* Depression exceeding mild depression (score > 19), as defined by Beck's Depression Inventory (BDI)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity change | Pain intensity at the beginning of the intervention and pain intensity change at 3 months and 12 months
  Measured by numeric rating scale (NRS) with a pain intensity ranging from "no pain" to "worst pain" (1 to 10) according to the conventional use of NRS

SECONDARY OUTCOMES:
Anxiety change | Anxiety at the beginning of the intervention and anxiety change at 3 months and 12 months.
  Anxiety symptoms are measured by State-Trait Anxiety Inventory (STAI)
Depression change | Depression at the beginning of the intervention and depression change at 3 months and 12 months.
  Depression is measured by Beck Depression Inventory (BDI), version II

CONTACTS AND LOCATIONS:
Overall Officials: Tage Orenius, Principal Investigator — Orton Orthopaedic Hospitla
Locations (1):
- Orton Orthopaedic Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orenius TI, Ristolainen L, Silen E, Hurri H. The Efficacy and Feasibility of an Interoceptive Exposure Technique for Preventing the Transition From Subacute to Chronic Back Pain by Altering the Emotional Response to Pain: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Oct 19;12:e45701. doi: 10.2196/45701. PMID 37856182